CLINICAL TRIAL: NCT02226614
Title: Development of a Head-cooling Device for Brain Injury: Healthy Volunteer Study
Brief Title: Development of a Head Cooling Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: vs1 25.03.14
Record Dates: First submitted 2014-07-22; First posted 2014-08-27 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2015-12

CONDITIONS: Body Temperature Changes
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- head cooling (Experimental): head cooling
  Interventions: Device: University of Edinburgh head cooling device

INTERVENTIONS:
Device: University of Edinburgh head cooling device — head cooling

SUMMARY:
This study is testing a head-cooling device on volunteers to assess temperature reduction.

ELIGIBILITY:
Inclusion Criteria:

* healthy humans

Exclusion Criteria:

* pregnant
* refusal of consent for registration with The Over-volunteering Protection Scheme

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Temperature change | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter Andrews, MD, Principal Investigator — University of Edinburgh
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom